CLINICAL TRIAL: NCT05024825
Title: Effect of Gabapentin on Postoperative Opioid Analgesic Use and Pain in Adolescents Undergoing Tonsillectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment target not met.
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Farzana Afroze, Assistant Professor of Anesthesiology, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4891
Record Dates: First submitted 2019-08-04; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative
Keywords: tonsillectomy; gabapentin; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Hydrocodone; Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): Patients in the gabapentin group will receive gabapentin preoperatively, one time dose of 10 mg/kg PO (maximum dose 600 mg) and will resume scheduled doses postoperatively of PO gabapentin, 300 mg PO every 8 hours, in addition to acetaminophen and ibuprofen for 7 days postoperative. Acetaminophen 15mg/kg PO (max 1 gm) every 4-6 hours as needed for pain, max dose 4 gm per day; Ibuprofen 4-10 mg/kg PO divided over 8 hours as needed for pain, max dose 40 mg/kg/day; gabapentin, 10 mg/kg standing every 8 hours (22).
  Interventions: Drug: Gabapentin
- Hydrocodone (Active Comparator): Patients in the hydrocodone group will receive scheduled doses of hydrocodone, acetaminophen and ibuprofen at scheduled doses. Acetaminophen 15mg/kg (max 1 gm) every 4-6 hours as needed for pain, max dose 4 gm per day; Ibuprofen 4-10 mg/kg PO divided over 8 hours as needed for pain, max dose 40 mg/kg/day; hydrocodone acetaminophen solution 7.5mg-325mg/15mL 5mL for ages 12-14yrs and 10 mL for ages 15-18yrs, q 4-6 hours as needed for pain.
  Interventions: Drug: hydrocodone, acetaminophen and ibuprofen

INTERVENTIONS:
Drug: Gabapentin — Patients in the gabapentin arm may at any point call the Pediatric ENT clinic if pain is not adequately controlled. Patients will be prescribed hydrocodone acetaminophen solution 7.5mg-325mg/15mL 5mL for ages 12-14 yrs and 10 mL for ages 15-18yrs, q 4-6 hours as needed for pain. Patients will be informed to stop taking gabapentin.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: hydrocodone, acetaminophen and ibuprofen — Patients in the hydrocodone group will receive scheduled doses of hydrocodone, acetaminophen and ibuprofen at scheduled doses. Acetaminophen 15mg/kg (max 1 gm) every 4-6 hours as needed for pain, max dose 4 gm per day; Ibuprofen 4-10 mg/kg PO divided over 8 hours as needed for pain, max dose 40 mg/kg/day; hydrocodone acetaminophen solution 7.5mg-325mg/15mL 5mL for ages 12-14yrs and 10 mL for ages 15-18yrs, q 4-6 hours as needed for pain.
  Other Names: no other intervention names applicable
  Arms: Hydrocodone

SUMMARY:
This study aims to determine if administration of gabapentin preoperatively followed by a standing postoperative course is effective in reducing and possibly eliminating the use of opioid analgesics following this procedure. As a secondary outcome, it will evaluate the possible improvement in post tonsillectomy pain control with the use of a standing dose of gabapentin.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded control trial designed to determine if administration of gabapentin postoperatively is effective in reducing and possibly eliminating the use of opioid analgesics following tonsillectomies in the adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12-18.
* Patient scheduled for elective tonsillectomy +/- adenoidec-tomy, +/- BMTs.
* ASA physical status I and II.

Exclusion Criteria:

* Severe upper respiratory tract infections.
* Patients who are actively on gabapentin or pregabalin, pre-existing with pain syndromes, chronic use of opioids, allergy to gabapentin, acetaminophen, and or NSAIDs
* Patient who lacks of fluency in English or inability to communicate pain.
* Patient who has severe asthma, bleeding disorders, and history of gastrointestinal bleeding, epilepsy, renal impairment or any other medical problem that in the opinion of the investigator would interfere with study population.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Total opioid equivalent dose | Through completion of the study. Time frame per subject is 7 days.
  The primary outcome variable will be the total opioid equivalent dose recorded over two weeks. The proposed study will test the null hypothesis that the two population (gabapentin and placebo) means are equal. The criterion for significance (alpha) has been set at 0.050. The test is 2-tailed, which means that an effect in either direction will be interpreted.

SECONDARY OUTCOMES:
Post operative pain score determined by Visual Analog Survey Scale | Through completion of the study. Time frame per subject is 7 days.
  Pain severity, The pain VAS is a unidimensional measure of pain intensity. Scale ranges from 1-10. Score of 0 indicates no pain. Score of 1-3 indicates mild pain, score of 4-6 indicates moderate pain, score of 6 is severe pain, score of 7-9 is very severe pain, and a score of 10 is worst pain possible.
Medication Adverse Effect | Through completion of the study. Time frame per subject is 7 days.
  Patient reported adverse effect to medications given

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Background] Fortuna RJ, Robbins BW, Caiola E, Joynt M, Halterman JS. Prescribing of controlled medications to adolescents and young adults in the United States. Pediatrics. 2010 Dec;126(6):1108-16. doi: 10.1542/peds.2010-0791. Epub 2010 Nov 29. PMID 21115581
- [Background] McCabe SE, West BT, Veliz P, McCabe VV, Stoddard SA, Boyd CJ. Trends in Medical and Nonmedical Use of Prescription Opioids Among US Adolescents: 1976-2015. Pediatrics. 2017 Apr;139(4):e20162387. doi: 10.1542/peds.2016-2387. Epub 2017 Mar 20. PMID 28320868
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update). Otolaryngol Head Neck Surg. 2019 Feb;160(1_suppl):S1-S42. doi: 10.1177/0194599818801757. PMID 30798778
- [Background] Crandall M, Lammers C, Senders C, Braun JV. Children's tonsillectomy experiences: influencing factors. J Child Health Care. 2009 Dec;13(4):308-21. doi: 10.1177/1367493509344821. Epub 2009 Oct 15. PMID 19833669
- [Background] Harley EH, Dattolo RA. Ibuprofen for tonsillectomy pain in children: efficacy and complications. Otolaryngol Head Neck Surg. 1998 Nov;119(5):492-6. doi: 10.1016/S0194-5998(98)70107-X. PMID 9807075
- [Background] Bedwell JR, Pierce M, Levy M, Shah RK. Ibuprofen with acetaminophen for postoperative pain control following tonsillectomy does not increase emergency department utilization. Otolaryngol Head Neck Surg. 2014 Dec;151(6):963-6. doi: 10.1177/0194599814549732. Epub 2014 Sep 9. PMID 25205639
- [Background] Hong SM, Cho JG, Chae SW, Lee HM, Woo JS. Coblation vs. Electrocautery Tonsillectomy: A Prospective Randomized Study Comparing Clinical Outcomes in Adolescents and Adults. Clin Exp Otorhinolaryngol. 2013 Jun;6(2):90-3. doi: 10.3342/ceo.2013.6.2.90. Epub 2013 Jun 14. PMID 23799166
- [Background] Haig GM, Bockbrader HN, Wesche DL, Boellner SW, Ouellet D, Brown RR, Randinitis EJ, Posvar EL. Single-dose gabapentin pharmacokinetics and safety in healthy infants and children. J Clin Pharmacol. 2001 May;41(5):507-14. doi: 10.1177/00912700122010384. PMID 11361047
- [Background] Sanders JG, Dawes PJ. Gabapentin for Perioperative Analgesia in Otorhinolaryngology-Head and Neck Surgery: Systematic Review. Otolaryngol Head Neck Surg. 2016 Dec;155(6):893-903. doi: 10.1177/0194599816659042. Epub 2016 Jul 26. PMID 27459955
- [Background] Hwang SH, Park IJ, Cho YJ, Jeong YM, Kang JM. The efficacy of gabapentin/pregabalin in improving pain after tonsillectomy: A meta-analysis. Laryngoscope. 2016 Feb;126(2):357-66. doi: 10.1002/lary.25636. Epub 2015 Sep 25. PMID 26404562
- [Background] Amani S, Abedinzadeh MR. Effects of Oral Gabapentin, Local Bupivacaine and Intravenous Pethidine on Post Tonsillectomy Pain. Iran J Otorhinolaryngol. 2015 Sep;27(82):343-8. PMID 26568937
- [Background] Retraction: Evaluation of gabapentin and dexamethasone alone or in combination for pain control after adenotonsillectomy in children. Saudi J Anaesth. 2018 Oct-Dec;12(4):662. doi: 10.4103/1658-354X.241421. PMID 30429763
- [Background] Yeganeh Mogadam A, Fazel MR, Parviz S. Comparison of analgesic effect between gabapentin and diclofenac on post-operative pain in patients undergoing tonsillectomy. Arch Trauma Res. 2012 Fall;1(3):108-11. doi: 10.5812/atr.7931. Epub 2012 Oct 14. PMID 24396757
- [Background] Amin SM, Amr YM. Comparison between preemptive gabapentin and paracetamol for pain control after adenotonsillectomy in children. Anesth Essays Res. 2011 Jul-Dec;5(2):167-70. doi: 10.4103/0259-1162.94758. PMID 25885382
- [Background] Moore A. Gabapentin and post tonsillectomy pain-the next best thing? Arch Trauma Res. 2013 Winter;1(4):188-90. doi: 10.5812/atr.9938. Epub 2013 Feb 1. No abstract available. PMID 24396778
- [Background] Jeon EJ, Park YS, Park SS, Lee SK, Kim DH. The effectiveness of gabapentin on post-tonsillectomy pain control. Eur Arch Otorhinolaryngol. 2009 Oct;266(10):1605-9. doi: 10.1007/s00405-008-0897-0. Epub 2008 Dec 20. PMID 19099314
- [Background] Mikkelsen S, Hilsted KL, Andersen PJ, Hjortso NC, Enggaard TP, Jorgensen DG, Hansen M, Henriksen J, Dahl JB. The effect of gabapentin on post-operative pain following tonsillectomy in adults. Acta Anaesthesiol Scand. 2006 Aug;50(7):809-15. doi: 10.1111/j.1399-6576.2006.01057.x. PMID 16879463
- [Background] Pande AC, Pollack MH, Crockatt J, Greiner M, Chouinard G, Lydiard RB, Taylor CB, Dager SR, Shiovitz T. Placebo-controlled study of gabapentin treatment of panic disorder. J Clin Psychopharmacol. 2000 Aug;20(4):467-71. doi: 10.1097/00004714-200008000-00011. PMID 10917408
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- See also: National Survey on Drug Use and Health: summary of national findings — https://www.samhsa.gov/data/sites/default/files/Revised2k11NSDUHSummNatFindings/Revised2k11NSDUHSummNatFindings/NSDUHresults2011.htm
- See also: National Vital Statistics System. Multiple cause of death file — https://www.cdc.gov/nchs/nvss/deaths.htm
- See also: Gabapentin Use in Postoperative and Neuropathic Pain in Children — https://med.virginia.edu/pediatrics/wp-content/uploads/sites/237/2015/12/Feb16_Gabapentin_PedPharmaco.pdf